CLINICAL TRIAL: NCT00720642
Title: Percutaneous Excision Trial (I-Pet): A Multi-Center Clinical Study Of The Intact Breast Lesion Excision System (Bles) To Demonstrate That A Definitive Diagnosis Can Be Made From The Tissue Sample Collected With The Intact Bles.
Brief Title: Percutaneous Excision Trial
Acronym: I-PET
Status: Completed | Type: Observational
Sponsor: Intact Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Intact 06-06
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Imaged Breast Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast lesion tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PSAP: This is the population of patients in whom surgical intervention could possibly be avoided. These patients will be those in whom all imaging evidence (mammographic or sonographic) was removed during the Intact BLES procedure, and in whom a definitive diagnosis of ADH could be made using the pathology assessment criteria outlined in the protocol.
- NPSAP: Patients with a pathology diagnosis of ADH in whom all imaging evidence (mammographic or sonographic) of the target lesion was NOT removed OR in whom a definitive diagnosis of ADH COULD NOT be made by implementing the pathology criteria for evaluation outlined in the protocol AND patients with a diagnosis of DCIS will undergo open surgical excision and will be analyzed separately from the PSAP group.

SUMMARY:
To confirm that a definitive diagnosis can be made from the tissue sample collected using the Intact BLES when defined radiology and pathology criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be a female at least 18 years of age at the time of Intact BLES biopsy
* Patient must have had an imaged abnormality found via mammography or sonography that warrants a biopsy for further diagnosis

Exclusion Criteria:

* Patients who have pre-pectoral breast implants
* Patients who have implantable devices such as pacemakers and defibrillators
* Patients who are pregnant or lactating
* Patients in whom the device is contraindicated
* Patients who are contraindicated for surgery due to factors such as anti-coagulant use which cannot be safely reversed or who exhibit fever or other clinical evidence of infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an imaged breast abnormality found with mammography or sonography whose initial biopsy will be taken with the Intact BLES.
Sampling Method: Non-Probability Sample
Enrollment: 1170 (Actual)
Dates: Start 2006-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients in various populations who undergo an Intact procedure with an upgrade in the diagnosis after undergoing an open surgical excision. | Post Intact Excision

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - University of Arkansas for Medical Services, Little Rock, Arkansas
  - The Breast Health Center, Indio, California
  - Long Beach Memorial Breast Center, Long Beach, California
  - The Hill Breast Center, Pasadena, California
  - Flagler Hospital, Saint Augustine, Florida
  - Center for Breast Care HCA, West Palm Beach, Florida
  - Metro Surgical Associates, Inc., Lithonia, Georgia
  - TIFT Regionald Medical Center, Tifton, Georgia
  - Maui Medical Group, Wailuku, Hawaii
  - Shawnee Mission Medical Center, Overland Park, Kansas
  - St. Joseph Medical Center, Towson, Maryland
  - Mercy Medical Center, Springfield, Massachusetts
  - Genesys Medical Center, Grand Blanc, Michigan
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Lourdes Hospital Breast Center, Binghamton, New York
  - Wilson Hospital Breast Center, Johnson City, New York
  - Jewish Hospital Breast Center, Cincinnati, Ohio
  - University of Cincinnati The Barrett Center, Cincinnati, Ohio
  - Elyria Memorial Hospital, Elyria, Ohio
  - St. John West Shore Hospital, Westlake, Ohio
  - Evangelical Hospital, Lewisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Coastal Carolina Breast Center, Murrells Inlet, South Carolina
  - Nashville Breast Center, Nashville, Tennessee